CLINICAL TRIAL: NCT01537159
Title: Quantitative DCE-MRI as a Predictor of Therapeutic Response in Acute Leukemia
Brief Title: MRI Assessment of Leukemia Response to Therapy
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Wei Huang, Associate Professor, OHSU Knight Cancer Institute
Other Study IDs: IRB00008123; HEM-11164-L (Other: OHSU Knight Cancer Institute); 8123 (Other: OHSU IRB)
Record Dates: First submitted 2012-02-14; First posted 2012-02-23 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Acute Myelogenous Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Myelogenous Leukemia (AML): Patients who have been diagnosed with AML
  Interventions: Device: 3 Tesla (3T) Siemens Total imaging matrix (TIM) Trio whole-body system

INTERVENTIONS:
Device: 3 Tesla (3T) Siemens Total imaging matrix (TIM) Trio whole-body system — Each MR scanning session will include the pre-contrast multi-slice T2-weighted MRI with fat-saturation and T1-weighted MRI which are regularly acquired in clinical protocols. Following these acquisitions, high-spatial and temporal-resolution DCE-MRI will be performed. The total duration of a research MR session is expected to be less than 45 min.
  Other Names: Magnetic Resonance Imaging (MRI)

SUMMARY:
The purpose of this study is to investigate if a type of magnetic resonance imaging (MRI) scan of the bone marrow before the start of standard chemotherapy can predict complete remission of leukemia patients after the therapy. This type of MRI scan, called dynamic contrast-enhanced MRI (DCE-MRI), measures bone marrow blood flow. For those patients who do not achieve complete remission status after initial therapy and will be treated with additional therapy, the investigators are also interested in determining if the second MRI exam before the additional therapy can predict complete remission. If successfully tested, the MRI exam may be used in the future to help with early identification of patients who are unlikely to respond to standard chemotherapy. This will allow for a personalized therapeutic plan to be developed for these patients at an early stage and prevent them from being exposed to toxic and ineffective therapies.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsed AML patients, who are scheduled to receive standard induction therapy.
* Age > 8 years and requiring no sedation.
* Patients must not be pregnant
* Women of childbearing potential must have negative serum pregnancy test performed within 7-days prior to start of study
* The subject or subject's legal guardian has the ability to understand and the willingness to sign a written informed consent and/or assent document. A signed study-specific informed consent and/or assent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Patients who would be normally excluded from undergoing an MRI examination - patients with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field.
* Patients who have known or suspected allergy to gadolinium-based contrast agent.
* Severe claustrophobia precluding subject from undergoing a MRI
* Patients with acute or chronic kidney dysfunction (estimated Glomerular Filtration Rate (eGFR) < 30ml/min/1.73 m2 as calculated using the Modification of Diet in Renal Disease (MDRD) Equation)
* Pregnant women are excluded from this study because of possible risk to the fetus.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Shutter-Speed Model | Up to 1 year
  To explore if Shutter-Speed Model (SSM) dynamic contrast-enhanced MRI (DCE-MRI)of the bone marrow (BM) can predict complete remission (CR) in newly diagnosed or relapsed acute myelogenous leukemia (AML)patients.

SECONDARY OUTCOMES:
Pilot Data | Up to 1 year
  To collect pilot data in SSM DCE-MRI assessment of AML response to therapy for the conduct of future studies.
Complete Response | Up to 1 year
  To explore whether SSM DCE-MRI differs in predicting complete response (CR) for the newly diagnosed AML patients and for the relapsed AML patients.
Second SSM DCE-MRI | Up to 1 year
  To explore if the second SSM DCE-MRI and/or changes between the first and second imaging studies can predict CR in the non-CR group who undergo an additional therapy.
DCE-MRI Biomarkers | Up to 1 year
  To compare/correlate/combine DCE-MRI bio-markers with micro-vascular density (MVD) and proangiogenic cytokine profiles for the purpose of predicting response of AML patients to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States